CLINICAL TRIAL: NCT04425707
Title: The Use of Ivermectin In the Treatment of COVID 19 Patients
Brief Title: Ivermectin In Treatment of COVID 19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, Dr. Ehab kamal, general director of fever hospitals, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-2020/3
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A ivermectin alone (Experimental): ivermectin will be administarted alone to COVID 19 patients
  Interventions: Drug: Ivermectin
- B standard care alone (Experimental): standard care will be administarted alone
  Interventions: Drug: Ivermectin
- C ivermectin added to standard of care (Active Comparator): ivermectin will be administarted in adition to standard care
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — use of Ivermectin in the treatment of COVID 19 patients, in comparison to and in addition to the standard care of treatment of COVID 19 in Egypt
  Other Names: hydroxychloroquine

SUMMARY:
as Egypt suffered a lot during the pandemic of COVID 19 with limited drug choices, many of the patients could not acheive viral clearence with the standard module of care teh idea of introduction of new medications in the treatment protocol of COVID 19 managment. Ivermectin had shown a promising results in vitro studies and in limited in vivo studies. this clinical trial may open a new hope for COVID 19 patients as a new and cheap line of treatment

DETAILED DESCRIPTION:
the study will compare the effect of ivermectin in comaprison and addition to the standard mode of care for the COVID 19 patients

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic mild cases and moderate cases proven to be infected by COVID 19 by viral RNA swap

Exclusion Criteria:

* Contraindications for the drug: hypersensitivity.
* Any medications with possible drug interactions.
* Severe cases.
* Any malignant condition.
* Pregnant females.
* Breast feeding females.
* Any patient on the following medications: Erdafitinib- Lasmiditan- Quinidine due to potential severe drug interaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
to evaluate the role of Ivermectin as a line of treatment for COVID 19 | 2 months
  the role of ivermectin in the cure of COVID 19 patients

SECONDARY OUTCOMES:
To asses the rate of viral clearance in comparison to other treatment protocols. | 2 months
  to compare the results of ivermectin with the standard care

CONTACTS AND LOCATIONS:
Overall Officials: houssam ho masoud, MD, Study Director — COVID sceintific comittee ministry of health and population
Locations (1):
- isolation and referal hospitals for COVID 19 patients, Cairo, Egypt